CLINICAL TRIAL: NCT00266929
Title: Comparing Surgical to Conservative Management in the Treatment of Type II Odontoid Fractures Among the Elderly
Brief Title: Treatment of Type II Odontoid Fractures Among the Elderly
Status: Completed | Type: Observational
Sponsor: AOSpine North America Research Network (Network)
Collaborators: AOSpine North America (Industry)
Responsible Party: Sponsor
Other Study IDs: 07-GOF-05
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Neck Injuries; Spinal Injuries
Keywords: odontoid fx; surgical intervention; conservative treatment; nonunion; odontoid fractures; surgical treatment
MeSH Terms: conditions — Neck Injuries; Spinal Injuries | interventions — Surgical Procedures, Operative; Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical: Subjects receiving surgical treatment for Type II odontoid fracture per discretion of investigator (non-randomized allocation)
  Interventions: Procedure: surgical
- Non-surgical: Subjects treated with non-operative treatment options
  Interventions: Procedure: conservative treatment

INTERVENTIONS:
Procedure: surgical — surgical treatment of odontoid fractures
  Groups: Surgical
Procedure: conservative treatment — conservative stabilization of fractures
  Groups: Non-surgical

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of surgical versus conservative management of type II odontoid fractures among patients > 64 years of age. Of secondary interest is to determine if there are differences in outcomes between anterior screw fixation and posterior fusion of these fractures.

DETAILED DESCRIPTION:
Hypotheses are as follows:

* Patients receiving surgical management will exhibit better disease specific health and general health related quality of life measures compared to those managed conservatively.
* The rate of radiographic bony fusion will be greater among elderly patients receiving surgical fixation compared to patients receiving conservative management.
* The rate of non union will be greater in the conservative group compared to the surgical group.
* The complication rate will be higher in the surgical group due to the nature of the intervention though the rate of severe and serious complications will be low.

ELIGIBILITY:
Inclusion Criteria:

* All new type II odontoid fractures including those in which the fracture line crosses into the body of C2
* Age > 64
* Stable and unstable fractures
* < 3 months post-injury
* No previous treatment for an odontoid fracture

Exclusion Criteria:

* Pathological fractures unrelated to osteoporosis
* Severe dementia or severe mental health problems
* Participation in other trials or unlikely to attend follow-ups

Min Age: 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects receiving care for acute Type II Odontoid Fracture in participating investigational sites
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2005-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Compare disease-specific health-related quality of life between the surgically and conservatively managed patients using the neck disability index | 12 months
Compare the proportion of patients with radiographic bony fusion between the surgically and conservatively managed patients | 12 months
Compare the rate of non-union between the surgically and conservatively managed patients | 12 months

SECONDARY OUTCOMES:
Compare the rate of complications | 12 months
Compare the cervical range of motion between patients receiving anterior screw fixation, posterior fusion, and conservative management | 12 months
Identify risk factors for a poor outcome, independent of treatment intervention | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander R Vaccaro, MD, Principal Investigator — Thomas Jefferson University and The Rothman Institute
Locations (15):
- United States (14):
  - Emory University SOM: Orthopedics, Atlanta, Georgia
  - Indiana Spine Group, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - John Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cornell Weill Medical College, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Spinal Cord Injury Center Thomas Jefferson University and The Rothman Institute, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Harborview Medical Center, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Smith HE, Kerr SM, Maltenfort M, Chaudhry S, Norton R, Albert TJ, Harrop J, Hilibrand AS, Anderson DG, Kopjar B, Brodke DS, Wang JC, Fehlings MG, Chapman JR, Patel A, Arnold PM, Vaccaro AR. Early complications of surgical versus conservative treatment of isolated type II odontoid fractures in octogenarians: a retrospective cohort study. J Spinal Disord Tech. 2008 Dec;21(8):535-9. doi: 10.1097/BSD.0b013e318163570b. PMID 19057244
- [Background] Smith HE, Vaccaro AR, Maltenfort M, Albert TJ, Hilibrand AS, Anderson DG, Harrop J, Fehlings MG, Kopjar B, Brodke DS, Arnold PM, Shaffrey CI. Trends in surgical management for type II odontoid fracture: 20 years of experience at a regional spinal cord injury center. Orthopedics. 2008 Jul;31(7):650. PMID 19292388
- [Result] Vaccaro AR, Kepler CK, Kopjar B, Chapman J, Shaffrey C, Arnold P, Gokaslan Z, Brodke D, France J, Dekutoski M, Sasso R, Yoon ST, Bono C, Harrop J, Fehlings MG. Functional and quality-of-life outcomes in geriatric patients with type-II dens fracture. J Bone Joint Surg Am. 2013 Apr 17;95(8):729-35. doi: 10.2106/JBJS.K.01636. PMID 23595072
- [Result] Fehlings MG, Arun R, Vaccaro AR, Arnold PM, Chapman JR, Kopjar B. Predictors of treatment outcomes in geriatric patients with odontoid fractures: AOSpine North America multi-centre prospective GOF study. Spine (Phila Pa 1976). 2013 May 15;38(11):881-6. doi: 10.1097/BRS.0b013e31828314ee. PMID 23459135
- [Result] Chapman J, Smith JS, Kopjar B, Vaccaro AR, Arnold P, Shaffrey CI, Fehlings MG. The AOSpine North America Geriatric Odontoid Fracture Mortality Study: a retrospective review of mortality outcomes for operative versus nonoperative treatment of 322 patients with long-term follow-up. Spine (Phila Pa 1976). 2013 Jun 1;38(13):1098-104. doi: 10.1097/BRS.0b013e318286f0cf. PMID 23354104
- [Result] Smith HE, Kerr SM, Fehlings MG, Chapman J, Maltenfort M, Zavlasky J, Harris E, Albert TJ, Harrop J, Hilibrand AS, Anderson DG, Vaccaro AR. Trends in epidemiology and management of type II odontoid fractures: 20-year experience at a model system spine injury tertiary referral center. J Spinal Disord Tech. 2010 Dec;23(8):501-5. doi: 10.1097/BSD.0b013e3181cc43c7. PMID 20940632
- [Result] Smith JS, Kepler CK, Kopjar B, Harrop JS, Arnold P, Chapman JR, Fehlings MG, Vaccaro AR, Shaffrey CI. Effect of type II odontoid fracture nonunion on outcome among elderly patients treated without surgery: based on the AOSpine North America geriatric odontoid fracture study. Spine (Phila Pa 1976). 2013 Dec 15;38(26):2240-6. doi: 10.1097/BRS.0000000000000009. PMID 24335630